CLINICAL TRIAL: NCT07037446
Title: A Multicenter, International, Prospective and Retrospective, Follow-up Registry to Monitor the Efficacy and Safety of the Occlutech Paravalvular Leak Device (PLD) in Patients With Mitral or Aortic Paravalvular Leaks
Acronym: PLD REGISTRY
Status: Enrolling by invitation | Type: Observational
Sponsor: Occlutech International AB (Industry)
Responsible Party: Sponsor
Other Study IDs: Occ2023_01
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-06

CONDITIONS: Paravalvular Leak Device (PLD)
Keywords: PLD Registry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Synopsis Title of the study A Multicenter, International, Prospective and Retrospective, Follow-up Registry to Monitor the Efficacy and Safety of the Occlutech Paravalvular Leak Device (PLD) in Patients with Mitral or Aortic Paravalvular Leaks Study Number Occ2023_01 Sponsor Occlutech International AB Landskronavägen 2 SE-252 32 Helsingborg Sweden Represented by Clinical Research Manager Gönül Sönmez Utkun Occlutech Tıbbi Urunler San.ve Tic.Ltd.Sti. Yeşilköy SB Mah. E Blok Sok, Occlutech Apt. No:6 34149, Istanbul, Turkey Coordinating Investigator Prof. Dr. Eustaquio Onorato, MD, FSCAI, FESC Unità Operativa di Cardiologia Universitaria Ospedale Galeazzi-Sant'Ambrogio, GSD, IRCCS Via Cristina Belgioioso, 173 20157 Milano, Italy Name of Investigational Device Occlutech® Paravalvular Leak Device (PLD) Indication The Occlutech PLD is a medical device intended to close a paravalvular leak (PVL). This leak is a relevant post-operational complication after the bioprosthetic or mechanical heart valve replacement or a result of paravalvular tissue rupture (early or late occurrence) or endocarditis, with possible lowintensity of heart murmurs. The PVL closure with the Occlutech PLD is indicated for patients with a significant leak that causes hemodynamically significant heart failure or hemolysis which requires recurrent blood transfusions.

It is further indicated for patients who are deemed at high risk for surgery after consultation with the surgeon or as an alternative to surgery with less operational time and recovery period.

Study purpose The objective of the study is to evaluate the safety and efficacy of the Occlutech PLD in patients requiring transcatheter closure of paravalvular leaks after previously implanted prosthetic heart valves. Study design This is an international, multicenter, retrospective and prospective, post marketing follow-up registry to monitor the efficacy and safety of the Occlutech® Paravalvular Leak Device (PLD) in subjects with mitral or aortic paravalvular leaks.

* Efficacy and safety of implanted device(s) will be assessed on Day 1 to 7, Day 30 (±15 days), 6 months to 1 year (±3 months), 1 year to 2 years (±3 months), 2 years to 3 years (±3 months) after the procedure.
* Patients will be treated according to the instruction-for-use of the device and according to clinical routine
* Procedures will be performed at sites having appropriate laboratory support and adequately trained interventional and imaging personnel. Procedure will be performed by physicians with experience in a wide range of interventional cardiology and structural heart disease, including transseptal puncture, anterograde, retrograde or transapical device delivery approaches to PVL interventions. Sample size consideration It is planned to enroll up to 200 subjects in which 150 subjects will be considered as evaluable subjects (i.e. followed-up for ≥1y) is a pragmatic approach for such a study, based on the recent publication of Onorato et al1. and 50 subjects are considered as drop-out (calculated as of 25% for the study). This guarantees 95%-CIs for continuous variables with a range of mean +/-0.16 standard deviations (SD), and binary variables (incidence or success rates r) with a range of r +/-0.16 (r(1 - r))½. This precision is sufficient for the descriptive study objective. Subject population Planned subject population: 200 subjects requiring transcatheter closure of paravalvular leaks after previously implanted prosthetic heart valves. Subjects will be screened to determine eligibility for this registry based on inclusion and exclusion criteria, medical history, demographic data, vital signs and clinical laboratory tests, ECG records and appropriate echocardiography. Study objectives
* To evaluate the safety of the Occlutech PLD by using its accessory and delivery system in patients requiring transcatheter closure of paravalvular leaks.
* To evaluate the efficacy of the Occlutech PLD by using its accessory and delivery system in patients requiring transcatheter closure of paravalvular leaks. Additional exploratory objectives To evaluate the compatibility and usability of the Occlutech PLD with the Occlutech Pistol Pusher (OPP) and the Occlutech Delivery Set III (ODS III) through a practitioner's questionnaire if applicable.

DETAILED DESCRIPTION:
Inclusion and Exclusion Criteria Inclusion Criteria

• Patient meeting the indication and area of application of the PLD device as described in the IFU.

The Occlutech® PLD is indicated for patients with a significant leak that causes hemodynamically significant heart failure or hemolysis which requires recurrent blood transfusions. It is further indicated for patients who are deemed at high risk for surgery or as an alternative to surgery after heart team evaluation including the surgeon.

* Male of female patients
* Patients of age ≥ 18 years
* Patients understanding the nature of the study and providing their informed consent to participation
* Patients willing and able to attend the follow-up visits and procedures foreseen by study CIP Exclusion Criteria

Contraindications as described in the IFU:

* Acute infection or any serious infection 1 month prior to procedure
* Adequate oral anti-coagulation therapy / platelet inhibition is not possible post-intervention
* Allergies to nickel and/or titanium and/or nickel/titanium-based materials Intolerance to contrast agents
* Known coagulation disorder
* Known intra-cardiac thrombus
* Recent pelvic venous thrombosis
* Recent myocardial infarction or a surgical bypass operation in the last 30 days NOTE: a positive result to a pregnancy test necessitates the exclusion of the subject from the registry. Study procedures Data will be collected using electronic case report forms (eCRF). Data collection will be based on clinical routine. Invasive assessments are optional and left to the discretion of the investigator.

NOTE: follow-up visits should be performed within the time windows as stated in Table 1.

Baseline data Patient's condition to qualify for this registry (refer to inclusion/exclusion criteria), date of informed consent. Demographics (age, gender) Medical history Relevant concomitant medication (name of medication, reason, dose, dose form, route of administration, frequency, start and date) Physical examination and vital signs (weight, height, NYHA Class, systolic/diastolic blood pressure, pulse rate, pregnancy test for female patients with childbearing potential) TTE/TEE/RT-2D/3D TEE (represents the best tool to assess the following parameters: number and position of the leaks, assessment of defect shape and size, regurgitation grade, LVEF, regurgitant volumes and fraction, VC, PHT, EDV, EROA) If needed for evaluation Multidetector Computed Tomography Angiography (MDCTA) / Cardiac Magnetic Resonance (CMR) Angiography (optional) (number and position of the leaks, assessment of defect shape and size, regurgitation grade, LVEF, regurgitant volumes and fraction) Electrocardiography (heart rate, sinus rhythm, atrial fibrillation, other arrhythmias) QoL Assessment Laboratory data (hematocrit, hemoglobin, LDH, iron, transferrine, ferritine, GFR, creatinine, urea, NT-proBNP), Number of hemolysis related blood transfusions Assessment and documentation of any new adverse events that may have occurred before implantation. Implantation / Post-procedure (Day 0) Device size and identification data (device reference number REF, device serial number SN, used accessory, accessory medical device serial number SN, accessory medical device reference number REF if there is more than one PVL, it's possible to implant devices following assessment should be performed accordingly) Implantation procedure (date, procedure-related complications, number of attempts for PVL(s) closure, duration, success/failure, type of echocardiography, fluoroscopy time, radiation dose) Assessment and documentation of any new or updated adverse events or adverse device effects that may have occurred after implantation and before discharge. Practitioner's Questionnaire for each accessory medical device used during the implantation will.be completed by Investigator (if applicable) Relevant concomitant medication (name of medication, reason, dose, dose form, route of administration, frequency, start and date) Follow-Up(1) at Day 1-7, Follow-Up(2) at 30 days (±15 days) , Follow-Up(3) at 6 months to 1 year (±3 months), Follow-Up(4) 1 - 2 years (±3 months), Follow- Up(5) 2-3 years (±3 months) after the procedure Physical examination and vital signs (weight, NYHA Class, systolic/diastolic blood pressure, pulse rate) TTE/TEE/RT-2D/3D TEE (represents the best tool to assess the following parameters: number and position of the leaks, assessment of defect shape and size, regurgitation grade, LVEF, regurgitant volumes and fraction, VC, PHT, EDV, EROA) If needed for evaluation If needed for evaluation Multidetector Computed Tomography Angiography (MDCTA) / Cardiac Magnetic Resonance (CMR) Angiography (optional) (number and position of the leaks, assessment of defect shape and size, regurgitation grade, LVEF, regurgitant volumes and fraction) Laboratory data (hematocrit, hemoglobin, LDH, NT-proBNP) Number of hemolysis related transfusions since last visit Assessment and documentation of any new or updated AEs/ADEs, SAEs/SADEs that may have occurred since implantation. Relevant concomitant medication (name of medication, reason, dose, dose form, route of administration, frequency, start and date) Electrocardiography (hearth rate, sinus rhythm, atrial fibrillation, other arrhythmias) Chest x-Ray (optional) QoL Assessment Data analysis and statistics Primary endpoint The primary safety endpoint is defined as the incidence of any Serious Adverse Device Effects (SADEs) including, but not limited to major cardiac arrhythmia (ventricular tachycardia/VF), procedure-related death, procedure-related stroke, rehospitalizations, systemic embolism, severe hemolysis, device embolization, infective endocarditis, prosthetic impingement, valvular regurgitation or vascular complications requiring surgery up to 1-year post-implantation, during the procedure new or worsening prothesis dysfunction, coronary obstruction, transfusion requirement, conversion to open surgery or unplanned intervention35 The primary efficacy endpoint is defined as successful implantation of the Occlutech PLD device with the recommended accessories and delivery system with effective closure of the paravalvular leak (defined as reduction in paravalvular regurgitation of ≥1 grade leak36 , presence of a residual PVL greater than mild as assessed by echocardiography post implantation) and reduction in the number of hemolysis-related transfusions assessed at 1-year post- implantation Follow-Up1,2.

Secondary endpoint Secondary safety endpoint is defined as the incidence of any Serious Adverse Device Effects (SADEs) including, but not limited to major cardiac arrhythmia (ventricular tachycardia/VF), procedure-related death, procedure-related stroke, acute kidney injury, systemic embolism, severe hemolysis, device embolization, infective endocarditis, prosthetic impingement, valvular regurgitation or bleeding/major vascular or cardiac structural complications requiring surgery from 1 year to 3-year post-implantation. This will also assess all minor complications such as transient hemolysis, vascular complications not requiring surgery, or all minor complications which are deemed relevant at the discretion of each investigator. Additionally, an assessment of all Serious Adverse Events (SAE) will be included in the analyses. Secondary efficacy endpoints refer to the variation in the data assessments from baseline to 3 years after the procedure in parameters such as, but not limited to, aortic blood pressure, pulse rate, LVFS, LDH, hematocrit, hemoglobin, regurgitation grade, NT-pro BNP value, ECG, NYHA classification and Quality of Life assessment1,2.

Secondary endpoints will be assessed:

* On day 1 to 7, Follow-Up 1
* At 30 days (±15 days), Follow-Up 2
* At 6 months to 1 year (±3 months), Follow-Up 3
* At 1-2 years (±3 months), Follow-Up 4
* At 2-3 years (±3 months), Follow-Up 5 after the procedure, following the Occlutech PLD device implantation. Additional exploratory endpoints The additional exploratory endpoint will assess the compatibility and usability of the Occlutech PLD device with the Occlutech Pistol Pusher (OPP) and the Occlutech Delivery Set (ODS) through a practitioner's questionnaire. Definition of population Full Analysis Set (safety and efficacy): All patients requiring treatment with the Occlutech PLD device, having at least one safety/efficacy assessment. Full Analysis Set (procedure): All patients belonging to the FAS (safety and efficacy), where treatment contains the accessory devices OPP and/or ODS III. Statistical analysis Continuous variables will be analyzed using descriptive statistics (numbers of observations and missing data, mean, standard deviation, median, minimum, maximum; categorical variables: frequency counts and percentages). For endpoints, two-sided 95%-confidence intervals will be reported in addition to the description.

For safety endpoints, besides the description of absolute and relative frequencies on the level of patients (patients with at least one event) and events, further statistical methods will be applied (evaluation of incidence rates). Details will be presented in the statistical analysis plan (SAP).

Interim analysis The sponsor reserves the right to perform a descriptive/administrative interim analysis at any time during the course of the registry. Safety Monitoring No additional burdensome or invasive procedures beyond the standard of care are requested by the investigational plan. However, an independent data and safety monitoring board is filed separately in the TMF. A final list will be shown in the clinical investigation / study report.

Data collection Data will be collected on electronic Case Report Forms (eCRFs). Study duration The maximum duration of each subjects' participation in this study is 3 years. It is planned to enroll up to 200 subjects in which 150 subjects will be considered as evaluable subjects (i.e. followed-up for ≥1y) is a pragmatic approach for such a study, based on the recent publication of Onorato et al.1 and 50 subjects are considered as drop-out (calculated as of 25% for the study).Based on the recent publication of Onorato et al.1 in which 144 subjects were enrolled in circa 6 years (21 sites in 10 countries), it is estimated that the planned number of subjects will be recruited within 4 years. As such, the estimated total duration of the study from first subject screened to last subject last visit is 7 years.

ELIGIBILITY:
Inclusion Criteria:

• Patient meeting the indication and area of application of the PLD device as laid down in the IFU.

The Occlutech® PLD is indicated for patients with a significant leak that causes hemodynamically significant heart failure or hemolysis which requires recurrent blood transfusions. It is further indicated for patients who are deemed at high risk for surgery after consultation with the surgeon or as an alternative to surgery with less operational time and recovery period.

* Male of female patients
* Patients of age ≥ 18 years
* Patients understanding the nature of the study and providing their informed consent to participation.
* Patients willing and able to attend the follow-up visits and procedures foreseen by study CIP.

Exclusion Criteria:

* Contraindications as described in the IFU:
* Acute infection or any serious infection 1 month prior to procedure
* Adequate oral anti-coagulation therapy / platelet inhibition is not possible post-intervention.
* Allergies to nickel and/or titanium and/or nickel/titanium-based materials
* Intolerance to contrast agents
* Known coagulation disorder
* Known intra-cardiac thrombus
* Recent pelvic venous thrombosis
* Recent myocardial infarction or a surgical bypass operation in the last 30 days Note: a positive result to a pregnancy test necessitates the exclusion of the subject from the registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Occlutech® PLD is indicated for patients with a significant leak that causes hemodynamically significant heart failure or hemolysis which requires recurrent blood transfusions. It is further indicated for patients who are deemed at high risk for surgery after consultation with the surgeon or as an alternative to surgery with less operational time and recovery period. The investigation population matches the target population.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | 1 year
  The primary safety endpoint is defined as the incidence of any Serious Adverse Device Effects (SADEs) including, but not limited to major cardiac arrhythmia (ventricular tachycardia/VF), procedure-related death, procedure-related stroke, rehospitalizations, systemic embolism, severe hemolysis, device embolization, infective endocarditis, prosthetic impingement, valvular regurgitation or vascular complications requiring surgery up to 1-year post-implantation, during the procedure new or worsening prothesis dysfunction, coronary obstruction, transfusion requirement, conversion to open surgery or unplanned intervention.

SECONDARY OUTCOMES:
Secondary endpoint | 3 year
  Secondary safety endpoint is defined as the incidence of any Serious Adverse Device Effects (SADEs) including, but not limited to major cardiac arrhythmia (ventricular tachycardia/VF), procedure-related death, procedure-related stroke, acute kidney injury, systemic embolism, severe hemolysis, device embolization, infective endocarditis, prosthetic impingement, valvular regurgitation or bleeding/major vascular or cardiac structural complications requiring surgery from 1 year to 3-year post-implantation. This will also assess all minor complications such as transient hemolysis, vascular complications not requiring surgery, or all minor complications which are deemed relevant at the discretion of each investigator. Additionally, an assessment of all Serious Adverse Events (SAE) will be included in the analyses.

CONTACTS AND LOCATIONS:
Locations (9):
- Turkey (Türkiye) (9):
  - İzmir Bayraklı Şehir Hastanesi, Izmir, Bayraklı
  - Gülhane Eğitim Araştırma Hastanesi, Ankara, Keçiören
  - Mehmet Akif Ersoy GKDC Eğitim Araştırma Hastanesi, Istanbul, Küçükçekmece
  - Tekirdağ Namık Kemal Üniversitesi Hastanesi, Tekirdağ, Süleymanpaşa
  - SBÜ Etlik Şehir Hastanesi Göğüs Kalp ve Damar Hastalıkları, Ankara, Yenimahalle
  - SBÜ Bursa Yüksek İhtisas Eğitim ve Araştırma Hastanesi, Bursa, Yıldırım
  - Hacettepe Üniversitesi, Ankara
  - Kocaeli Üniversitesi Hastanesi, Kocaeli
  - Özel Ankara Güven Hastanesi, Ankara, Çankaya